CLINICAL TRIAL: NCT00040222
Title: Clinical, Genetic, Behavioral, Laboratory and Epidemiologic Characterization of Individuals and Families at High Risk of Breast/Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020212; 02-C-0212; NCT00045214 (obsolete NCT alias)
Record Dates: First submitted 2002-06-22; First posted 2002-06-24 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-06-27

CONDITIONS: Familial Ovarian Cancer; Familial Breast Cancer; BRCA1-associate Malignancies; BRCA2-associated Malignancies
Keywords: Counseling/behavioral/psychosocial; Gene discovery; Cancer prevention; Risk-reduction; Hereditary; Natural History; Breast Cancer; Ovarian Cancer; Cowden Syndrome; Peutz-Jegher Syndrome; Li-Fraumeni Syndrome
MeSH Terms: conditions — Breast Cancer, Familial; Risk Reduction Behavior; Breast Neoplasms; Ovarian Neoplasms; Hamartoma Syndrome, Multiple; Peutz-Jeghers Syndrome; Li-Fraumeni Syndrome

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Individuals and families with known or suspected syndromes that include breast, ovarian or genetically-related cancers are enrolled in this family study.

SUMMARY:
Individuals and families with known or suspected syndromes that include breast, ovarian or genetically-related cancers are enrolled in this family study, which is a syndrome-specific sub-set of the long-standing DCEG Human Genetics Program umbrella family studies protocol (78-C-0039). Cancer outcomes are documented through review of medical, vital, and pathology records. Selected individuals and family members are asked to complete questionnaires to assess etiologic risk factors and to undergo clinical evaluations specifically tailored to the relevant familial syndrome. Study participants are monitored prospectively for the development of outcomes of interest, typically by means of periodic mail or telephone contact. In selected instances, subjects may return to the Clinical Center periodically for study-specific follow-up examinations. Study participants are asked to donate biologic specimens to be used in the laboratory search for cancer etiology and mechanisms of carcinogenesis. DNA and serial serum samples will be collected. Tumor tissue will be obtained whenever feasible.

Clinical genetic testing for tumor susceptibility gene(s) mutations and risk notification will be offered consistent with ASCO guidelines when reasonable individual cancer risk estimates can be delivered, and only to those participants who choose to know their individual genetic status after appropriate education and counseling. The testing will be conducted exclusively in Clinical Laboratory Improvement Amendments (CLIA)-licensed laboratories. Clinical genetic testing and risk notification are entirely optional and do not affect subject eligibility for other aspects of the protocol. A separate consent procedure and consent form will be used for genetic testing and risk notification.

This protocol, developed in response to recommendations developed by the Clinical Center IRB, is intended to:

1. Provide a mechanism under which the Clinical Genetics Branch can honor the commitment made to the members of over 60 hereditary breast/ovarian cancer families which have been participated in various Human Genetics Program research studies conducted over the past 3 decades to provide genetic counseling,

   clinical germline mutation testing, and consultative services now that several of the major breast/ovarian cancer susceptibility genes have been identified;
2. Provide a mechanism through which new families with various familial syndromes associated with an increased risk of breast and ovarian cancer can be studied, as research interests in these syndromes evolve over time; and
3. Create a resource of well-characterized, carefully documented high-risk families to facilitate the development of new etiologic and translational research studies in the future.

While we do not offer specific anti-cancer therapy as part of this protocol, we provide assistance to ensure that study participants who require treatment for problems that develop during the course of the study are referred to appropriate health providers. We

remain available to provide advice and consultation related to the management of the familial cancer syndrome to study participants and their health care providers.

DETAILED DESCRIPTION:
Individuals and families with known or suspected syndromes that include breast, ovarian or genetically-related cancers are enrolled in this family study, which is a syndrome-specific sub-set of the long-standing DCEG Human Genetics Program umbrella family studies protocol (78-C-0039). Cancer outcomes are documented through review of medical, vital, and pathology records. Selected individuals and family members are asked to complete questionnaires to assess etiologic risk factors and to undergo clinical evaluations specifically tailored to the relevant familial syndrome. Study participants are monitored prospectively for the development of outcomes of interest, typically by means of periodic mail or telephone contact. In selected instances, subjects may return to the Clinical Center periodically for study-specific follow-up examinations. Study participants are asked to donate biologic specimens to be used in the laboratory search for cancer etiology and mechanisms of carcinogenesis. DNA and serial serum samples will be collected. Tumor tissue will be obtained whenever feasible.

Clinical genetic testing for tumor susceptibility gene(s) mutations and risk notification will be offered consistent with ASCO guidelines when reasonable individual cancer risk estimates can be delivered, and only to those participants who choose to know their individual genetic status after appropriate education and counseling. The testing will be conducted exclusively in Clinical Laboratory Improvement Amendments (CLIA)-licensed laboratories. Clinical genetic testing and risk notification are entirely optional and do not affect subject eligibility for other aspects of the protocol. A separate consent procedure and consent form will be used for genetic testing and risk notification.

This protocol, developed in response to recommendations developed by the Clinical Center IRB, is intended to:

1. Provide a mechanism under which the Clinical Genetics Branch can honor the commitment made to the members of over 60 hereditary breast/ovarian cancer families which have been participated in various Human Genetics Program research studies conducted over the past 3 decades to provide genetic counseling, clinical germline mutation testing, and consultative services now that several of the major breast/ovarian cancer susceptibility genes have been identified;
2. Provide a mechanism through which new families with various familial syndromes associated with an increased risk of breast and ovarian cancer can be studied, as research interests in these syndromes evolve over time; and
3. Create a resource of well-characterized, carefully documented high-risk families to facilitate the development of new etiologic and translational research studies in the future.

While we do not offer specific anti-cancer therapy as part of this protocol, we provide assistance to ensure that study participants who require treatment for problems that develop during the course of the study are referred to appropriate health providers. We remain available to provide advice and consultation related to the management of the familial cancer syndrome to study participants and their health care providers.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals age 18 and over are considered for inclusion in the study if they have a:

Family history of neoplasia of an unusual type, pattern, or number which includes breast cancer or is consistent with an identified or suspected familial cancer syndrome which includes breast and/or ovarian cancer,

Personal history of neoplasia(s) or benign conditions of an unusual type or with unusual demographic features (young age of onset, multiple primary sites, rare tumor type of pathologic characteristics) consistent with an identified or suspected familial cancer syndrome which includes breast and/or ovarian cancer, or

A known mutation associated with one of the breast/ovarian cancer family syndromes.

Eligibility is now restricted to only bloodline individuals age 18 and over from families which are already enrolled in 02-C-0212 and in which there is a known BRCA mutation

Personal and family medical history must be verified through questionnaires, interviews, and review of pathology slides and medical records. For known or suspected familial syndromes in which no gene has been identified, two or more living affected cases among family members are required for participation. The types of familial syndromes under active accrual and study are predominantly investigator-and hypothesis-driven. This approach permits CGB investigators to remain alert to the opportunities afforded by unexpected clusters of rare tumors in families and individuals, and to tailor the accrual of families with specific types of syndromes to meet programmatic goals. This requires that CGB investigators remain abreast of both general knowledge and state-of the-art developments in clinical oncology, genetics, epidemiology and molecular biology, so that critical research opportunities can be recognized when they present, and so that thoughtful decisions can be made regarding the commitment of the resources needed to conduct such studies.

EXCLUSION CRITERIA:

Individuals and families referred for evaluation in whom reported diagnoses are not verifiable.

Inability to provide informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals and families with known or suspected syndromes that include breast, ovarian or genetically-related cancers are enrolled in this family study.
Sampling Method: Non-Probability Sample
Enrollment: 377 (Actual)
Dates: Start 2002-07-01 (Actual)

PRIMARY OUTCOMES:
Epidemiologic Characterization of Individuals and Families at High Risk of Breast/Ovarian Cancer | Ongoing
  To ascertain individuals and families at high risk of breast, ovarian andother syndromically related cancers due to known or suspected genetic factor(s) which predispose to neoplasia in order to:- Evaluate and define the clinical spectrum and natural history of disease in syndromes predisposing to familial breast/ovarian cancer;- Develop a resource of epidemiologic, clinical, behavioral and genetic information on individuals and families predisposed to familial breast/ovarian cancer; - Track and validate cancer occurrence and other clinical outcomes in members of these highrisk kindreds;- Create a biospecimen repository which will facilitate exploratory,etiologically-focused laboratory studies;- Evaluate potential precursor states of neoplastic disease in families atrisk of breast and ovarian cancer;- Quantify the risk of specific tumors in family members;- Map, clone, and determine the function of novel tumor susceptibilitygenes
Genetic and Environmental Factors | Ongoing
  Identify genetic determinants, and genetic and environmental modifiers of cancer risk in individuals and families predisposed tobreast/ovarian cancer; and- Evaluate gene-gene and gene-environment interactions in thepathogenesis of familial breast/ovarian cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon A Savage, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bojesen SE, Pooley KA, Johnatty SE, Beesley J, Michailidou K, Tyrer JP, Edwards SL, Pickett HA, Shen HC, Smart CE, Hillman KM, Mai PL, Lawrenson K, Stutz MD, Lu Y, Karevan R, Woods N, Johnston RL, French JD, Chen X, Weischer M, Nielsen SF, Maranian MJ, Ghoussaini M, Ahmed S, Baynes C, Bolla MK, Wang Q, Dennis J, McGuffog L, Barrowdale D, Lee A, Healey S, Lush M, Tessier DC, Vincent D, Bacot F; Australian Cancer Study; Australian Ovarian Cancer Study; Kathleen Cuningham Foundation Consortium for Research into Familial Breast Cancer (kConFab); Gene Environment Interaction and Breast Cancer (GENICA); Swedish Breast Cancer Study (SWE-BRCA); Hereditary Breast and Ovarian Cancer Research Group Netherlands (HEBON); Epidemiological study of BRCA1 & BRCA2 Mutation Carriers (EMBRACE); Genetic Modifiers of Cancer Risk in BRCA1/2 Mutation Carriers (GEMO); Vergote I, Lambrechts S, Despierre E, Risch HA, Gonzalez-Neira A, Rossing MA, Pita G, Doherty JA, Alvarez N, Larson MC, Fridley BL, Schoof N, Chang-Claude J, Cicek MS, Peto J, Kalli KR, Broeks A, Armasu SM, Schmidt MK, Braaf LM, Winterhoff B, Nevanlinna H, Konecny GE, Lambrechts D, Rogmann L, Guenel P, Teoman A, Milne RL, Garcia JJ, Cox A, Shridhar V, Burwinkel B, Marme F, Hein R, Sawyer EJ, Haiman CA, Wang-Gohrke S, Andrulis IL, Moysich KB, Hopper JL, Odunsi K, Lindblom A, Giles GG, Brenner H, Simard J, Lurie G, Fasching PA, Carney ME, Radice P, Wilkens LR, Swerdlow A, Goodman MT, Brauch H, Garcia-Closas M, Hillemanns P, Winqvist R, Durst M, Devilee P, Runnebaum I, Jakubowska A, Lubinski J, Mannermaa A, Butzow R, Bogdanova NV, Dork T, Pelttari LM, Zheng W, Leminen A, Anton-Culver H, Bunker CH, Kristensen V, Ness RB, Muir K, Edwards R, Meindl A, Heitz F, Matsuo K, du Bois A, Wu AH, Harter P, Teo SH, Schwaab I, Shu XO, Blot W, Hosono S, Kang D, Nakanishi T, Hartman M, Yatabe Y, Hamann U, Karlan BY, Sangrajrang S, Kjaer SK, Gaborieau V, Jensen A, Eccles D, Hogdall E, Shen CY, Brown J, Woo YL, Shah M, Azmi MA, Luben R, Omar SZ, Czene K, Vierkant RA, Nordestgaard BG, Flyger H, Vachon C, Olson JE, Wang X, Levine DA, Rudolph A, Weber RP, Flesch-Janys D, Iversen E, Nickels S, Schildkraut JM, Silva Idos S, Cramer DW, Gibson L, Terry KL, Fletcher O, Vitonis AF, van der Schoot CE, Poole EM, Hogervorst FB, Tworoger SS, Liu J, Bandera EV, Li J, Olson SH, Humphreys K, Orlow I, Blomqvist C, Rodriguez-Rodriguez L, Aittomaki K, Salvesen HB, Muranen TA, Wik E, Brouwers B, Krakstad C, Wauters E, Halle MK, Wildiers H, Kiemeney LA, Mulot C, Aben KK, Laurent-Puig P, Altena AM, Truong T, Massuger LF, Benitez J, Pejovic T, Perez JI, Hoatlin M, Zamora MP, Cook LS, Balasubramanian SP, Kelemen LE, Schneeweiss A, Le ND, Sohn C, Brooks-Wilson A, Tomlinson I, Kerin MJ, Miller N, Cybulski C, Henderson BE, Menkiszak J, Schumacher F, Wentzensen N, Le Marchand L, Yang HP, Mulligan AM, Glendon G, Engelholm SA, Knight JA, Hogdall CK, Apicella C, Gore M, Tsimiklis H, Song H, Southey MC, Jager A, den Ouweland AM, Brown R, Martens JW, Flanagan JM, Kriege M, Paul J, Margolin S, Siddiqui N, Severi G, Whittemore AS, Baglietto L, McGuire V, Stegmaier C, Sieh W, Muller H, Arndt V, Labreche F, Gao YT, Goldberg MS, Yang G, Dumont M, McLaughlin JR, Hartmann A, Ekici AB, Beckmann MW, Phelan CM, Lux MP, Permuth-Wey J, Peissel B, Sellers TA, Ficarazzi F, Barile M, Ziogas A, Ashworth A, Gentry-Maharaj A, Jones M, Ramus SJ, Orr N, Menon U, Pearce CL, Bruning T, Pike MC, Ko YD, Lissowska J, Figueroa J, Kupryjanczyk J, Chanock SJ, Dansonka-Mieszkowska A, Jukkola-Vuorinen A, Rzepecka IK, Pylkas K, Bidzinski M, Kauppila S, Hollestelle A, Seynaeve C, Tollenaar RA, Durda K, Jaworska K, Hartikainen JM, Kosma VM, Kataja V, Antonenkova NN, Long J, Shrubsole M, Deming-Halverson S, Lophatananon A, Siriwanarangsan P, Stewart-Brown S, Ditsch N, Lichtner P, Schmutzler RK, Ito H, Iwata H, Tajima K, Tseng CC, Stram DO, van den Berg D, Yip CH, Ikram MK, Teh YC, Cai H, Lu W, Signorello LB, Cai Q, Noh DY, Yoo KY, Miao H, Iau PT, Teo YY, McKay J, Shapiro C, Ademuyiwa F, Fountzilas G, Hsiung CN, Yu JC, Hou MF, Healey CS, Luccarini C, Peock S, Stoppa-Lyonnet D, Peterlongo P, Rebbeck TR, Piedmonte M, Singer CF, Friedman E, Thomassen M, Offit K, Hansen TV, Neuhausen SL, Szabo CI, Blanco I, Garber J, Narod SA, Weitzel JN, Montagna M, Olah E, Godwin AK, Yannoukakos D, Goldgar DE, Caldes T, Imyanitov EN, Tihomirova L, Arun BK, Campbell I, Mensenkamp AR, van Asperen CJ, van Roozendaal KE, Meijers-Heijboer H, Collee JM, Oosterwijk JC, Hooning MJ, Rookus MA, van der Luijt RB, Os TA, Evans DG, Frost D, Fineberg E, Barwell J, Walker L, Kennedy MJ, Platte R, Davidson R, Ellis SD, Cole T, Bressac-de Paillerets B, Buecher B, Damiola F, Faivre L, Frenay M, Sinilnikova OM, Caron O, Giraud S, Mazoyer S, Bonadona V, Caux-Moncoutier V, Toloczko-Grabarek A, Gronwald J, Byrski T, Spurdle AB, Bonanni B, Zaffaroni D, Giannini G, Bernard L, Dolcetti R, Manoukian S, Arnold N, Engel C, Deissler H, Rhiem K, Niederacher D, Plendl H, Sutter C, Wappenschmidt B, Borg A, Melin B, Rantala J, Soller M, Nathanson KL, Domchek SM, Rodriguez GC, Salani R, Kaulich DG, Tea MK, Paluch SS, Laitman Y, Skytte AB, Kruse TA, Jensen UB, Robson M, Gerdes AM, Ejlertsen B, Foretova L, Savage SA, Lester J, Soucy P, Kuchenbaecker KB, Olswold C, Cunningham JM, Slager S, Pankratz VS, Dicks E, Lakhani SR, Couch FJ, Hall P, Monteiro AN, Gayther SA, Pharoah PD, Reddel RR, Goode EL, Greene MH, Easton DF, Berchuck A, Antoniou AC, Chenevix-Trench G, Dunning AM. Multiple independent variants at the TERT locus are associated with telomere length and risks of breast and ovarian cancer. Nat Genet. 2013 Apr;45(4):371-84, 384e1-2. doi: 10.1038/ng.2566. PMID 23535731
- [Background] Kramer JL, Velazquez IA, Chen BE, Rosenberg PS, Struewing JP, Greene MH. Prophylactic oophorectomy reduces breast cancer penetrance during prospective, long-term follow-up of BRCA1 mutation carriers. J Clin Oncol. 2005 Dec 1;23(34):8629-35. doi: 10.1200/JCO.2005.02.9199. PMID 16314625
- [Background] Loud JT, Gierach GL, Veenstra TD, Falk RT, Nichols K, Guttmann A, Xu X, Greene MH, Gail MH. Circulating estrogens and estrogens within the breast among postmenopausal BRCA1/2 mutation carriers. Breast Cancer Res Treat. 2014 Feb;143(3):517-29. doi: 10.1007/s10549-013-2821-6. Epub 2014 Jan 18. PMID 24442642
- [Derived] Korde LA, Mueller CM, Loud JT, Struewing JP, Nichols K, Greene MH, Mai PL. No evidence of excess breast cancer risk among mutation-negative women from BRCA mutation-positive families. Breast Cancer Res Treat. 2011 Jan;125(1):169-73. doi: 10.1007/s10549-010-0923-y. Epub 2010 May 11. PMID 20458532
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2002-C-0212.html